CLINICAL TRIAL: NCT04130906
Title: A Feasibility Trial of Theta Burst Stimulation in Binge Eating Disorder
Brief Title: Theta Burst Stimulation in Binge Eating Disorder: A Single Session RCT
Acronym: BITE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID led to suspension of the study.New data suggest outcome measures should be revised and new approvals from research ethics committees will be needed.
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pending
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Binge-Eating Disorder
Keywords: Binge Eating; Transcranial Magnetic Stimulation; Theta Burst Stimulation; Neuromodulation; Psychiatric Disorders; Eating Disorders
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Mental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Theta Burst Stimulation (Active Comparator): The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer active iTBS.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Sham Intermittent Theta Burst Stimulation (Sham Comparator): The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer TBS using a sham Magstim coil.
  Interventions: Device: Sham Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — iTBS will be delivered to the left dorsolateral prefrontal cortex (DLPFC) at 80% of resting motor threshold using standard stimulation parameters; triplet-bursts will be delivered at high frequency (50 Hz) with an inter-burst interval of 200 ms. Each TBS train will last 2 seconds and consists of 10 triplet-bursts (30 pulses). Each iTBS session will involve 10 TBS trains repeated every 10 seconds for 190 seconds, with a total number of 600 pulses delivered during each session.
  Other Names: iTBS
  Arms: Intermittent Theta Burst Stimulation
Device: Sham Intermittent Theta Burst Stimulation — Sham stimulation will be delivered left dorsolateral prefrontal cortex (DLPFC) using the same parameters as real iTBS however, a sham coil will be used. The sham coil makes the same noise and creates a similar sensation on the scalp as the real coil but does not produce a magnetic field.
  Other Names: Sham TBS
  Arms: Sham Intermittent Theta Burst Stimulation

SUMMARY:
Binge eating disorder (BED) is a common and disabling eating disorder (ED) which presents a substantial disease burden. Individuals seeking treatment for binge eating difficulties typically receive talking therapy treatment however, treatment response is inadequate. As such, it is imperative that novel treatment options be identified.

Repetitive transcranial magnetic stimulation (rTMS) techniques are well established for the treatment of depression and preliminary findings indicate that similarly therapeutic effects may occur in populations with eating difficulties. Intermittent theta burst stimulation (iTBS) is a novel variant of excitatory rTMS which is emerging as an attractive alternative to standard stimulation. This trial aims to assess the feasibility of conducting a large scale randomised controlled trial (RCT) investigating theta burst in individuals with binge eating disorder, and to examine whether theta burst stimulation may improve symptoms in this population.

DETAILED DESCRIPTION:
Binge eating is a common and disabling problem which is often associated with obesity. Binge eating causes significant distress and compromises quality of life in affected individuals. To date current treatments do not support full recovery in a considerable number of adults and adolescents. As such, it is important that we explore new options for treatment.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive procedure that is emerging as a potentially effective treatment for a range of psychiatric disorders. In rTMS, an electric current is passed through a coil placed on the scalp. This current creates a magnetic field which changes the activity in the brain area immediately below the coil. rTMS is a well-established treatment for depression and has been approved by the National Institute for Care and Excellence (NICE; 2015). The NICE-approved rTMS treatment for depression involves 20-30 sessions, each requiring 37.5 minutes of stimulation. A novel variant of rTMS, intermittent theta burst stimulation (iTBS), is an attractive alternative to standard stimulation; TBS, which is delivered using a very similar procedure as standard rTMS, may produce effects comparable to standard rTMS in as little as 3 minutes.

In depression, the therapeutic applications for rTMS have been widely studied. By comparison, research examining the potential applications of rTMS for the treatment of eating disorders and obesity are preliminary. Nevertheless, studies in eating disorders and obesity to date have reported promising results. For example, a case study involving a patient with refractory BED and comorbid depression reported clinical improvement following 20 sessions of high frequency (excitatory) rTMS targeting the left DLPFC (Baczynski et al, 2014). Similarly, two recent studies of obese adults have reported a reduction in food intake, reduced craving, and significant weight loss following 20 sessions of high frequency rTMS targeting the left DLPFC (Alvarado-Reynoso & Ambriz-Tututi, 2019; Kim et al, 2018). Finally, studies in healthy participants reporting strong cravings and clinical participants with bulimia nervosa have also reported a reduction in craving and food-intake following high frequency rTMS (for example, Dunlop et al, 2015; Van den Eynde, 2010, and Uher et al, 2010). No study to date has used iTBS in eating disorders.

The primary objective for this trial is to assess whether iTBS may benefit people with binge eating difficulties. As such, we are conducting two inter-related studies: (1) a proof-of-concept randomised double-blind sham-controlled trial involving a single-session of either real or sham iTBS, and (2) a therapeutic case series involving 20 sessions of real iTBS delivered week-daily over four consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Meets DSM-5 criteria for full-syndrome BED
* Overweight or obese according to World Health Organisation (WHO) criteria (BMI>25 kg/m2 for adults, and a weight-for-height greater than 2 standard deviations above the median for adolescents).

Exclusion Criteria:

* All known contraindications to MRI and TBS (assessed using TMS and MRI safety screening questionnaires)
* Pregnancy (or suspected pregnancy)
* History of neurological disease and/or seizure
* Having any metallic implants anywhere in the head or body
* History of head or eye injury; significant health problems in the previous six months;
* Lifetime diagnosis of substance dependence, psychosis, bipolar disorder, borderline personality disorder
* Other primary psychiatric disorder requiring treatment in its own right
* Taking psychotropic medication other than a stable dosage of selective serotonin reuptake inhibitors (SSRI) for at least 14 days prior to study enrollment
* Alcohol consumption exceeding 14 units per week
* Cigarette consumption or nicotine replacement exceeding >15 cigarettes daily or equivalent.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Binge Eating Disorder Visual Analogue Scale Measure of Symptom Severity | Baseline, within 1 hour after receiving active or sham stimulation, and 24-hour follow-up
  An index of BED symptoms will be computed by summing the scores on four 10cm visual analogue scales (VAS) assessing levels of current hunger, craving for food, urge to eat and urge to binge eat. Participants will indicate along the line the extent to which they are experiencing the symptom described, with a mark at 0cm indicating "None" and 10cm indicating "Extreme". Higher scores indicate higher BED severity.

SECONDARY OUTCOMES:
Visual Analogue Scale Measure of General Psychopathology | Baseline, within 1 hour after receiving active or sham stimulation, and 24-hour follow-up
  An index of "related psychopathology" will be computed by summing the scores on four 10cm visual analogue scales (VAS) assessing feeling low, level of tension, level of stress and level of anxiety will then be completed. Participants will indicate along the line the extent to which they are experiencing the symptom described, with a mark at 0cm indicating "None" and 10cm indicating "Extreme". Higher scores indicate greater symptom severity.
Delay Discounting Task | Baseline, within 1 hour after receiving active or sham stimulation, and 24-hour follow-up
  Participants complete a series of 27 questions that each require choosing between a smaller, immediate reward (e.g., £25 today) versus a larger, later reward (e.g., £35 in 25 days). Modeling techniques are used to fit the function that relates time to discounting. The main dependent measure of interest is the change in the steepness of the discounting curve from baseline to post-iTBS; A more steeply declining curve represents a tendency to devalue rewards as they become more temporally remote (i.e., further way).
Emotion Regulation Task | Baseline, within 1 hour after receiving active or sham stimulation, and 24-hour follow-up
  Participants will view images from the international affective picture schedule and be asked to either experience their emotions naturally or to use a reappraisal strategy to increase or decrease their emotional experience. Heart rate data will be collected during task completion. The main dependent measure of interest is change in high frequency heart rate variability for each condition (watch or reappraise) from baseline to post TBS.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schmidt, Principal Investigator — King's College London
Locations (1):
- King's College London Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No